CLINICAL TRIAL: NCT06590350
Title: Individualized NUTRItional RISK and Oriented Nutritional Support
Acronym: NUTRISKO
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6407 - NUTRISKO
Record Dates: First submitted 2024-03-29; First posted 2024-09-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort who received clinical nutrition counseling <72 hours: Patients at risk of malnutrition who received clinical nutrition counseling within 72 hours.
  Interventions: Other: Clinical nutrition counseling
- Cohort who did NOT received clinical nutrition counseling <72 hours: Patients at risk of malnutrition who did NOT receive clinical nutrition counseling within 72 hours.
  Interventions: Other: Clinical nutrition counseling

INTERVENTIONS:
Other: Clinical nutrition counseling — In the first phase, all patients admitted to the Departmental Simple Operating Unit Admission Room of Policlinico Universitario A. Gemelli will be screened for NRS-2002 upon admission.
  Only patients with NRS-2002 ≥ 3 will subsequently be tracked via the Foundation's computer system (TrackCare®).
  The patients will be managed by caregivers who may spontaneously request nutritional counseling, as is currently the case.
  Patient data (laboratory tests, medical history, reason for admission, any instrumental test reports) and clinical outcomes (average length of hospitalization, complications, antibiotic therapy use, intensive care admission, mortality, re-hospitalization within 30 days) will be obtained from the Foundation's computer system (TrackCare®) and recorded in a dedicated Excel® spreadsheet.
  Costs related to hospitalization and management of any complications will also be assessed.

SUMMARY:
The objective of this study is to evaluate whether, in patients who are given early nutritional counseling, there is a reduction in the length of hospitalization and the rate of nosocomial infections, resulting in a decrease in inpatient costs, compared with patients who do not benefit from this intervention.

DETAILED DESCRIPTION:
Patients admitted from the date following the date of approval of the protocol for the following 12 months will be enrolled at the Departmental Simple Operating Unit Admission Room of the Policlinico Universitario A. Gemelli and who have undergone NRS-2002 screening.

Data only of patients with NRS-2002 > 3 admitted will be considered and extracted via the Foundation's computer system (Trackcare).

Patients will be managed by caregivers who spontaneously request (as is the case to date) nutritional counseling. Therefore, the study will not change current clinical practice.

Two cohorts will be formed and compared:

Cohort 1: patients at risk of malnutrition (NRS-2002 ≥ 3) who received clinical nutrition counseling within 72 hours of ward admission.

Cohort 2: patients at risk of malnutrition (NRS-2002 ≥ 3) who did NOT receive clinical nutrition counseling beyond 72 hours after ward admission.

Currently, at Fondazione Policlinico Universitario A. Gemelli, the Clinical Nutrition Unit is approached on an ad hoc basis by the individual ward attending physician, without a specific procedure: the physician calls in Clinical Nutrition specialists for consultation if in his or her judgment the patient needs nutritional support. The formation of the two cohorts will be entirely spontaneous, that is, according to current clinical practice, given by the judgment of the ward treating physician. In a spontaneous manner, two cohorts will be formed among patients at risk of malnutrition (NRS-2002 ≥ 3), one of which will have received specialized nutritional support within 72 hours, the other will not. Only patients at risk of malnutrition will be tracked, highlighting outcomes among those in this category who received the targeted intervention at the appropriate times, versus those who did not. The enrollment department is the same for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* NRS-2002 ≥3
* Length of stay > 4 days
* Informed consent to participate in the study

Exclusion Criteria:

* NRS-2002 <3
* Length of stay < or = 4 days
* Absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at risk of malnutrition by default (NRS-2002 ≥3) admitted to the Admission Room Departmental Simple Operating Unit of the A. Gemelli Polyclinic Foundation in Rome.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Difference in the duration of hospitalization | 12 months
  Difference in the overall length of stay in patients at risk of malnutrition (NRS-2002 ≥ 3) who received nutrition counseling within 72 hours of ward admission compared to the group of patients at risk who did not receive counseling within 72 hours.

SECONDARY OUTCOMES:
Differences in the number of infectious complications | 12 months
  Difference in the overall length of stay in patients at risk of malnutrition (NRS-2002 ≥ 3) who received nutrition counseling within 72 hours of ward admission compared to the group of patients at risk who did not receive counseling within 72 hours.
Frequency of adherence to diet and AFMS proposed at visit | 12 months
  requency of adherence to the prescribed diet and AFMS (Artificial Feeding and Medical Support) proposed during the visit.
Differences in hospitalization costs for the healthcare | 12 months
  Differences in hospitalization costs for the healthcare facility among patients at risk of malnutrition who received nutritional counseling within 72 hours of admission compared to the group of patients at risk who did not receive counseling within 72 hours of ward entry.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Rinninella, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Emanuele Rinninella, Rome, Italy